CLINICAL TRIAL: NCT00316875
Title: A Phase I, Open-Label Study of the Safety, Tolerability and Pharmacokinetics of Lapatinib in Combination With Liposomal Doxorubicin in Patients With Metastatic Breast Cancer
Brief Title: Lapatinib and Doxorubicin Hydrochloride Liposome in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, William Gradishar, Principal Investigator, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 05B5; P30CA060553 (NIH); NU-05B5; NU-1838-001; NCI-2011-00325 (Other: NCI CTRP#)
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Lapatinib; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lapatinib Ditosylate and Doxil (Experimental)
  Interventions: Drug: lapatinib ditosylate; Drug: Doxil

INTERVENTIONS:
Drug: lapatinib ditosylate — 1500 mg orally daily for as long as patients remain on trial (up to 8 cycles).
Drug: Doxil — Administered intravenously (IV) every 4 weeks in a dose-escalating fashion according to a set schedule
  Other Names: Doxorubicin HCL Liposome Injection; Dox-SL

SUMMARY:
RATIONALE: Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as doxorubicin hydrochloride liposome work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving lapatinib together with doxorubicin hydrochloride liposome may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of doxorubicin hydrochloride liposome when given together with lapatinib in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the safety, tolerability, and feasibility of pegylated doxorubicin HCl liposome (PLD) when administered with lapatinib, particularly in terms of cardiac safety, in patients with metastatic breast cancer.
* Determine the optimally tolerated regimen (OTR) of PLD when administered with lapatinib in these patients.

Secondary

* Determine the pharmacokinetic profiles of lapatinib and PLD when given in combination at the OTR.
* Describe any preliminary evidence of efficacy of lapatinib and PLD in these patients.

OUTLINE: This is an open-label, dose-escalation study of pegylated doxorubicin HCl liposome (PLD).

Patients receive oral lapatinib once daily on days 1-28 and PLD IV over at least 30 minutes on day 1. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Lapatinib may be continued alone in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of PLD until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 6 patients experience dose-limiting toxicity.

After completing study treatment, patients are followed for 30 days.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast with evidence of metastatic disease

  * Epidermal growth factor receptor (EGFR) and/or erbB2 positivity not required
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension as ≥ 20 mm by conventional techniques OR as ≥ 10 mm by spiral CT scan
* No known brain metastases or leptomeningeal disease
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Male or female patients
* Menopausal status not specified
* Life expectancy ≥ 12 weeks
* ECOG performance status 0-1
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin normal
* AST/ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* LVEF ≥ 50%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow and retain oral medication
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to lapatinib
* No gastrointestinal (GI) tract disease resulting in inability to take oral medication
* No malabsorption syndrome or requirement for IV alimentation
* No uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis)

PRIOR CONCURRENT THERAPY:

* Prior trastuzumab (Herceptin ®) allowed
* Prior anthracyclines allowed provided total dose of doxorubicin hydrochloride ≤ 240 mg/m² or epirubicin ≤ 600 mg/m²
* More than 4 weeks since prior major surgery, hormonal therapy (other than replacement therapy), chemotherapy (6 weeks for nitrosoureas or mitomycin C), or radiotherapy and recovered
* No prior surgical procedures affecting absorption
* No prior EGFR-targeting therapies
* At least 7 days since prior and no concurrent CYP3A4 inhibitors
* At least 7 days since prior and no concurrent gastric pH modifiers

  * Antacids allowed within 1 hour before and after lapatinib dosing
* At least 14 days since prior and no concurrent CYP3A4 inducers, including dexamethasone or dexamethasone equivalent dose > 1.5 mg/day
* At least 6 months since prior and no concurrent amiodarone
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent prophylactic growth factor support
* No concurrent herbal medications
* No other concurrent investigational agents or anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Cardiac safety | Throughout treatment and up to 30 days post-treatment
Maximum tolerated dose | After the first cycle of therapy

SECONDARY OUTCOMES:
Pharmacokinetic profiles | After treatment completion for 12 patients treated at the maximum tolerated dose
Efficacy | At time of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: William J Gradishar, M.D., Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States